CLINICAL TRIAL: NCT06053385
Title: Impact of Commercial "Sleep Lotion" on Salivary Melatonin Levels and Sleep Quality in Undergraduates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Redlands (Other)
Responsible Party: Principal Investigator, Lisa Olson, Professor of Biology, University of Redlands
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2021-37-REDLANDS
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sleep
Keywords: melatonin; lotion

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the melatonin lotion first or the placebo control lotion first, and then each participant will receive the other treatment second.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin sleep lotion Night 1; Placebo control lotion Night 2 (Experimental): Participants in this arm received melatonin-containing "sleep lotion" to apply on the first night of saliva sampling. On the second night of saliva sampling, they received placebo control lotion.
  Interventions: Other: Melatonin sleep lotion; Other: Placebo control lotion
- Placebo control lotion Night 1; Melatonin sleep lotion Night 2 (Experimental): Participants in this arm received placebo control lotion to apply on the first night of saliva sampling. On the second night of saliva sampling, they received melatonin-containing "sleep lotion."
  Interventions: Other: Melatonin sleep lotion; Other: Placebo control lotion

INTERVENTIONS:
Other: Melatonin sleep lotion — 7 g of lotion applied to hands and arms one hour before bedtime
  Other Names: Dr. Teal's Sleep Lotion
Other: Placebo control lotion — 7 g of lotion applied to hands and arms one hour before bedtime
  Other Names: Dr. Teal's Lavender Essential Oils Lotion

SUMMARY:
The goal of this clinical trial is to test an over-the-counter "sleep lotion" in healthy undergraduate college students. The main questions it aims to answer are:

* Does an over-the-counter "sleep lotion" containing melatonin actually increase melatonin levels in participants compared to a placebo (control) lotion?
* Does an over-the-counter "sleep lotion" containing melatonin improve the quality of participants' sleep compared to a placebo (control) lotion?

Participants will:

* provide three saliva samples on each of two nights
* apply melatonin-containing "sleep lotion" on one night and a placebo (control with no melatonin) lotion on the other night
* answer questionnaires about gender, race, ethnicity, medication use, exercise, and sleep quality

DETAILED DESCRIPTION:
Melatonin is a hormone secreted by the pineal gland in the brain that regulates sleep. There are many over-the-counter products such as bubble baths, room sprays, and lotions that claim they contain melatonin and promote sleep. This study is a randomized, controlled, double-blind crossover trial to compare the impact of a commercial "sleep lotion" vs. a control lotion on melatonin levels detectable in saliva in healthy undergraduate students. Participants will provide saliva samples on two nights, one week apart, one hour before bedtime. The sample collections will take place just before and twice after applying 1) a melatonin lotion and 2) a placebo control lotion (order randomized). The investigators will determine whether the melatonin lotion affects the natural rise of melatonin before bedtime. A second dependent variable will be the quality of sleep on both nights. Potential confounding independent variables, such as gender, race, ethnicity, medication use, and exercise will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 24 years old
* current University of Redlands student

Exclusion Criteria:

* Pregnancy
* currently taking any sleep medications
* allergies or sensitivities to scented lotion

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Salivary melatonin | Three samples over an hour: pre-lotion application (one hour before bedtime), 30 minutes after lotion application, and one hour after lotion application (at bedtime). This 1 hr sampling will happen on two separate nights within a week of enrollment.
  pg/ml of melatonin in saliva measured by enzyme-linked immunosorbent assay
Sleep Quality | A 15 minute questionnaire taken each morning after lotion application and saliva sampling. These two mornings are both within a week of enrollment (specific dates chosen by participant).
  Modified Pittsburgh Sleep Quality Index. Scores from 0 (good sleep quality) to 14 (poor sleep quality)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Olson, Ph.D., Principal Investigator — University of Redlands
Locations (1):
- University of Redlands, Redlands, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be provided upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting after publication, and up to 10 years after publication
Access Criteria: Will be provided to researchers affiliated with an academic institution upon request

REFERENCES:
- [Derived] Ponce C, Razon AD, Chao J, Nakagawa SK, Peterson MM, Roque AY, Vanderpool MA, Ferracane MJ, Olson LE. Impact of an over-the-counter "sleep lotion" on human salivary melatonin levels and sleep quality: a randomized controlled trial. Neuro Endocrinol Lett. 2024 Aug 12;45(3):167-172. PMID 39146562